CLINICAL TRIAL: NCT04156399
Title: Acupuncture for Adults With Sickle Cell Disease (SCD): A Feasibility Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the Coronavirus Disease 2019 (COVID-19) pandemic
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Judith Schlaeger, Assistant Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-1077
Record Dates: First submitted 2019-11-01; First posted 2019-11-07 (Actual); Results first posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-02

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; pain; chronic pain; acupuncture
MeSH Terms: conditions — Anemia, Sickle Cell; Pain; Chronic Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: This study is an unblinded, uncontrolled trial.
Masking Description: There is no masking. This study is unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acupuncture (Experimental): All subjects will receive active acupuncture.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — All subjects will receive a standardized 18 needle acupuncture protocol.

SUMMARY:
The investigators long-term goal is to demonstrate the effectiveness of acupuncture for the treatment of adults with chronic pain due to sickle cell disease (SCD), a debilitating pain syndrome characterized by acute and chronic pain. The objective of this study is to explore the feasibility and acceptability of acupuncture with adult patients with SCD. All participants will receive acupuncture treatments twice per week for 5 weeks. Subjects will complete measures at baseline and post-treatment, and a measure of study acceptability at post-treatment. The investigators will describe the procedures and potential challenges to implementing the acupuncture protocol, and expect to identify and rectify any procedural problems that subjects report regarding the 10-session study protocol.

DETAILED DESCRIPTION:
The investigators will conduct the study with adults with chronic pain from SCD, 18 years old or greater. They will all receive acupuncture. Treatments will be twice weekly for 5 weeks, for 30 minutes per treatment. At baseline and post-treatment, subjects will complete measures that include pain, fatigue, anxiety, depressive symptoms, injustice experience, and pain catastrophizing. Subjects will also complete a measure of study acceptability, the Protocol Acceptability Scale for Treating SCD with Acupuncture at post-treatment. The investigators will describe the procedures and potential challenges to implementing the acupuncture protocol and the range in the subjects' Acceptability Scale scores. The investigators will expect to identify and rectify any procedural problems that subjects will report regarding the 10-session study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adults with Sickle Cell Disease
* Receiving care at the University of Illinois Sickle Cell Disease clinic
* Moderate to severe level of pain (3 or higher on a 0-10 scale) within the last 3 months

Exclusion Criteria:

* Pregnancy
* Physically or cognitively unable to complete the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith M Schlaeger, PhD, Principal Investigator — UIC
Locations (1):
- University of Illinois at Chicago College of Nursing, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li H, Patil CL, Molokie RE, Njoku F, Steffen AD, Doorenbos AZ, Schlaeger JM. Acupuncture for chronic pain in adults with sickle cell disease: a mixed-methods pilot study. Acupunct Med. 2021 Dec;39(6):612-618. doi: 10.1177/09645284211017303. Epub 2021 Jun 3. PMID 34080441

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acupuncture
Started | 6
Completed | 2 (Of the six participants who started the study, two completed all 10 acupuncture sessions, two completed 9 sessions, and one completed 8 sessions. The three who completed 8 or 9 sessions were unable to complete due to the COVID-19 lockdowns, however, we were able to collect post-test measures for them. Finally, one participant was hospitalized (unrelated to acupuncture) and could not complete the study nor provide post-test measures.)
Not Completed | 4
Not completed — hospitalization unrelated to acupuncture | 1
Not completed — study suspension due to COVID pandemic | 3

BASELINE CHARACTERISTICS:
Arm/Group | Acupuncture
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Performing Acupuncture for the Treatment of Chronic Pain in Adults With SCD.
Description: Feasibility was measured in terms of participant enrollment and retention and participant completion of study measures. The investigators screened 9 potential participants of which 6 were found to be eligible and all 6 consented to participate and started the study (100% recruitment of eligible SCD patients). Of the 6, 2 completed 10 treatments; 3 completed 8 or 9 treatments by the time the coronavirus disease 2019 (COVID-19) started, but had not missed any treatments and would have most likely completed if the study had not been halted, and completed all pre and post measures (83% retention). The 6th person could not complete because she was hospitalized, but probably would have completed otherwise.
  Feasibility and acceptability were the only pre-specified outcome measures.
Time Frame: After 10th acupuncture treatment, at 5 weeks post-baseline (study completion)
Measure: Number; unit: participants
Arm/Group | Acupuncture
Number analyzed (Participants) | 5
participants
  Potential participants eligible | 6
  Participants consented/started study | 6
  Participants completed | 5
  Participants not completed | 1

2. Primary Outcome: Protocol Acceptability Scale for Treating Sickle Cell Disease With Acupuncture
Description: Protocol Acceptability Scale for Treating SCD with Acupuncture is a 10-item instrument with scores ranging from 0 to 20 used to measure acceptability of the study processes and protocols. Items are measured on a 0 to 2 scale, where 0 means "did not like the study/did not like acupuncture/did not enjoy participating", and 2 means "liked the study/liked acupuncture/enjoyed participating". The protocol was deemed to have high acceptability if 80% of participants scored ≥ 80% of possible points on the acceptability scale. The investigators calculated the mean score for each of the 10 questions, divided the total score for the 10 questions by the maximum possible points for the measure, and converted the total mean scores to percentage of participants who liked the study/liked acupuncture/enjoyed participating.
  Feasibility & acceptability were the specified outcome measures.
Time Frame: After 10th acupuncture treatment, at 5 weeks post-baseline (study completion)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acupuncture
Number analyzed (Participants) | 5
score on a scale | 16.4 (2.8)

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
A limitation of the study is that it had to be terminated early due to COVID-19 lockdowns, resulting in only 6 recruited and 5 participants analyzed. Another limitation is the inability to complete all acupuncture sessions on 3 participants due to the pandemic. In addition, the one-armed design reduced the ability to test significant changes in measures (pain intensity, pain interference, fatigue, sleep disturbance, depression, anxiety, and anger) before and after the acupuncture intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT04156399/Prot_SAP_000.pdf